CLINICAL TRIAL: NCT04133779
Title: Multiple Sclerosis
Brief Title: Observational Study on Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Fondazione Italiana Sclerosi Multipla (Other)
Responsible Party: Sponsor
Other Study IDs: FondazioneISM
Record Dates: First submitted 2019-10-04; First posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Health Records, Personal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Group A (MS): * Age 18-55 years;
  * Unisex patients diagnosed with MS according to McDonald criteria and successive relapse (38, 39), and subjects with CIS;
  * Course of the disease: RR-SP-PP-CIS;
  * Disease duration (starting from diagnosis): from 1 month to 25 years for subjects with RR, SP, and PP; a maximum of 5 years for subjects with CIS;
  * Not in clinical relapse (at least 30 days after the last clinical relapse);
  * Subjects treated or non-treated with immunomodulatory and immunosupressive drugs;
  * Signature of the informed consent.
  Interventions: Procedure: neurological examination, Kurtzke EDSS, Barthel scale, ecocolor-Doppler
- Group B (HC): * Age 18-55 years;
  * Absence of significant diseases and lack of familiarity with MS, ie health check-ups (HC);
  * Signature of the informed consent.
  The subjects included in this group could be, for example, unrelated relatives or spouses of those affected by MS or other diseases in the study, or linked to these by affinity restrictions (such as, the father-in-law with the son-in-law, the husband with his wife's brother, etc.) or accompanying persons or operators of other centres.
  Interventions: Procedure: medical history, vital signs, ecocolor-Doppler
- Group C (OND): * Aged 18-55 years;
  * Subjects with other non-inflammatory neurodegenerative disease (OND), for example Parkinson, ALS, ataxy.
  * Signature of the informed consent.
  Interventions: Procedure: neurological evaluation, ecocolor-Doppler
- Group D (ONDi): * Age 18-55 years;
  * subjects suffering of other inflammatory neurodegenerative diseases (ONDi), for example optical neuromielitys, ADEM, encephalitis, neuro lupus, neurological complications of systemic autoimmune diseases;
  * Signature of the informed consent.
  Interventions: Procedure: neurological evaluation, ecocolor-Doppler

INTERVENTIONS:
Procedure: neurological examination, Kurtzke EDSS, Barthel scale, ecocolor-Doppler — For the subjects diagnosed with MS (group A), who did not need to be in a period of clinical relapse of the disease (at least 30 days from the last clinical relapse), the duration and the form of the disease was indicated (CIS, RR, SP or PP). The Investigator has submitted these subjects to a neurological examination which included the standard neurological examination, the Kurtzke EDSS (Kurtzke Expanded Disability Status Scale) comprising the functional systems of Kurtzke and the Barthel scale. After completing the selection phase following the previous examinations, the subjects were directed towards the qualified practitioner for the ecocolor-Doppler examination which was performed in blind.
  Groups: Group A (MS)
Procedure: neurological evaluation, ecocolor-Doppler — For the subjects affected by OND and ONDi, as in the groups C and D respectively, the Investigator has performed, beside the anamnesis and the physical examination, a specific neurological evaluation which included the compilation of the Barthel scale for the disability evaluation. After completing the selection phase following the previous examinations, the subjects were directed towards the qualified practitioner for performing the ecocolor-Doppler examination which was performed in blind.
  Groups: Group C (OND); Group D (ONDi)
Procedure: medical history, vital signs, ecocolor-Doppler — For the healthy subjects (HC) of the group B, the Investigator has solely performed the medical history and a check of the vital signs, reporting the demographic and clinical data of the subjects. After completing the selection phase following the previous examinations, the subjects were directed towards the qualified practitioner for the ecocolor-Doppler examination which was performed in blind.
  Groups: Group B (HC)

SUMMARY:
This is a multicentre observational study which involves 43 of the major Italian centres that treat MS. The duration expected for the study participation of each subject was exclusively the necessary one for the screening visit and execution of the ecocolor-Doppler test, which could have also been executed on the same day.

ELIGIBILITY:
Inclusion Criteria:

* Group A (MS)

  * Age 18-55 years;
  * Unisex patients diagnosed with MS according to McDonald criteria and successive relapse (38, 39), and subjects with CIS;
  * Course of the disease: RR-SP-PP-CIS;
  * Disease duration (starting from diagnosis): from 1 month to 25 years for subjects with RR, SP, and PP; a maximum of 5 years for subjects with CIS;
  * Not in clinical relapse (at least 30 days after the last clinical relapse);
  * Subjects treated or non-treated with immunomodulatory and immunosuppressive drugs;
  * Signature of the informed consent.

Group B (HC)

* Age 18-55 years;
* Absence of significant diseases and lack of familiarity with MS, ie health check-ups (HC);
* Signature of the informed consent.

The subjects included in this group could be, for example, unrelated relatives or spouses of those affected by MS or other diseases in the study or linked to these by affinity restrictions (such as, the father-in-law with the son-in-law, the husband with his wife's brother, etc.) or accompanying persons or operators of other centres.

Group C (OND)

* Aged 18-55 years;
* Subjects with other non-inflammatory neurodegenerative disease (OND), for example Parkinson, ALS, ataxy.

Group D (ONDi)

* Age 18-55 years;
* subjects suffering of other inflammatory neurodegenerative diseases (ONDi), for example optical neuromielitys, ADEM, encephalitis, neuro lupus, neurological complications of systemic autoimmune diseases;
* Signature of the informed consent.

Exclusion Criteria:

* • The presence of acute or chronic disease which are disabling or interfere with the design and objective of the study;

  * Clinically proven cardiopathy (NYHA ≥ I class);
  * Previous episodes of venal thromboembolism (including either deep venal thrombosis or pulmonary embolism);
  * Neoplasms;
  * Thrombophilia from an anamnestic definition;
  * Diabetes;
  * Primary or secondary pulmonary hypertension and in treatment for it;
  * Concurrent systemic steroid treatments or in the last 30 days;
  * Cerebrovascular diseases current or previous;
  * Episodes of global transitory amnesia;
  * Pregnancy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects aged 18-55 years, non-gender based, non-sex based.
Sampling Method: Probability Sample
Enrollment: 1767 (Actual)
Dates: Start 2010-12-29 (Actual); Primary Completion 2012-05-30 (Actual); Study Completion 2012-05-30 (Actual)

PRIMARY OUTCOMES:
The presence of CCSVI | 29.12.2010-30.05.2012
  The protocol provided that the presence of CCSVI was evaluated according to the Zamboni criteria at local level. Therefore, the ecocolor-Doppler images were sent in a randomized process to a central assessor who performed the first centralized reading. In case of disagreement with the local reading, the same images were to be sent to other two central readers, preserving the anonymity, in order to obtain a final evaluation in regards to the CCSVI presence.

IPD SHARING:
Plan to Share IPD: Undecided